## **Document Coversheet**

Study Title: Exploring an Incubator to Decrease Stress in Farmers Occupational Stress and Depression in Beginning Kentucky Farmers

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 3/7/22 |
| NCT Number: | NCT04932018 |
| IRB Number | 61320 |
| Coversheet created: | 11/15/22 |



IRB Approval 3/7/2022 IRB # 61320 IRB3

751 Rose Street 315 College of Nursing Lexington, KY 40536-0232

U

## Dear Kentucky farmer:

Researchers at the University of Kentucky are inviting you to take part in a 6-month research study about your experiences as a beginning farmer, depression, and your occupational stress "farm stress" level. The title of the study is: "Exploring the feasibility of a start-up incubator to decrease occupational stress and depression in beginning Kentucky farmers." The purpose of this study is to determine the feasibility of a start-up incubator intervention designed to decrease occupational stress and depression for beginning Kentucky farmers. The objectives are to: #1) test the feasibility of a mentorship and start-up incubator intervention on depression in beginning Kentucky farmers using questionnaires administered prestudy, mid-study, and post-study; #2) explore associations between mentorship, occupational stress and depression in beginning Kentucky farmers using specific survey questionnaires to guide future research. This study's results will provide valuable data to agriculture and occupational health researchers. The data will illustrate the impact of mentorship and community support on improving depression and occupational stress of beginning Kentucky farmers.

This study consists of electronic surveys that are being offered to beginning Kentucky farmers (by the USDA definition and live in any county in Kentucky. After identifying your eligibility, you will have a link to the survey and you will be assigned to one of two groups and we will ask that you do the following: **Group A** will participate at least once monthly in an online virtual community and complete online survey OR **Group B** will participate at least once monthly in an online virtual community and complete online survey PLUS

- 1. <u>Baseline:</u> complete <u>one</u> electronic survey at the beginning of the study
- <u>2. Second timepoint: complete one electronic survey at the mid-point of the study:</u>
- 3. Third time point: complete one electronic survey at the end of the study, **plus** Group B will attend an in-person meeting. Supper will be served at this meeting. Date to be determined.

Participation in this research study is voluntary. There are no known risks associated with participation in this study. Although you may not get personal benefit from taking part in this research study, your responses will help us understand more about beginning farmers, occupational stress and depression. Some volunteers experience satisfaction from knowing they have contributed to research that may possibly benefit others in the future. The surveys will take approximately 20 minutes to complete; participation in the virtual community will take less than 1 hour; and the in-person meeting (Group B) will take approximately 2 hours. Group A will be given a novelty t-shirt and access to the virtual community for 1 year for taking part in this study; Group B will also receive supper provided at the in-person meeting. The only costs associated with participation in this study is the cost of transportation to the in-person dinner for Group B, held in your county of residence. All participants will receive a \$20 Wal-Mart gift card upon enrollment in the study. Your response to the survey is confidential which means no names will appear or be used on research documents or be used in presentations or publications. The PI will communicate with all participants via email or in the virtual community designed specifically for this study protocol. All information obtained during this study will be stored in a secure location accessible only to the principal investigator and study coordinator. Please be aware, while we make every effort to safeguard your data once received on our servers via REDCap, given the nature of online surveys, as with anything involving the Internet, we can never guarantee the confidentiality of online data while in route to us. At the end of the study, all records will be destroyed after 6 years. We hope to receive completed questionnaires from about 48 people, so your answers are important to us. Of course, you have a choice about whether to complete the survey questionnaires or not, but if you do participate, you are free to skip any questions or discontinue at any time. If you do not want to be in the study, there are no other choices except to not take part in the study. If you have questions about the study, please feel free to ask; my contact information is given below. If you have complaints, suggestions, or questions about your rights as a research volunteer, contact the staff in the University of Kentucky Office of Research Integrity at 859-257-9428 or toll-free at 1-866-400-9428.

LINK TO SURVEY: https://redcap.uky.edu/redcap/surveys/?s=JJ9TJN3HND

Thank you in advance for your assistance in this important project. To ensure your responses will be included, submit your completed survey as soon as possible.

Sincerely,

John

College of Nursing, University of Kentucky

Phone: 859-323-0639

Martin & Brade

Julie Derringer, MSN RN CEN

Occupation and Environmental Health Nursing Trainee

PhD Student, University of Kentucky

Phone: 502-382-6568

